CLINICAL TRIAL: NCT03046134
Title: Burden of Hospitalized Pneumonia and Its Clinical Characteristics in Korea COPD Population: A Prospective, Multi-center, Cohort Study
Brief Title: Burden of Hospitalized Pneumonia in Korea COPD Population
Acronym: COPDCAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, JAE YEOL KIM, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Other Study IDs: WI221325
Record Dates: First submitted 2017-02-01; First posted 2017-02-08 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: COPD; Pneumonia; Pneumococcal Vaccine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: PCV13 — Conjugated pneumococcal vaccine

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the leading causes of morbidity and mortality worldwide. By 2030, COPD is expected to be the fourth main cause of death. Community-acquired pneumonia (CAP) represents not only a frequent complication but also a deadly cause in COPD patients. Inhaled corticosteroids, which are frequently used among COPD patients increase the risk for pneumonia. The effect of pneumococcal conjugate vaccine 13 (PCV13) on the prevention of pneumococcal pneumonia among COPD patients in Korean population has not been studied yet.

Several factors such as multi-lobar pneumonia, Pseudomonas aeruginosa pneumonia, and high pneumonia severity are related to poor outcome of patients with COPD and pneumonia. Prior pneumococcal vaccine has a beneficial effect on outcomes of pneumonia with COPD patients. However, the effects of pneumococcal vaccine on the clinical outcome of COPD patients were evaluated mainly on 23-valent pneumococcal polysaccharide vaccine (PPV23). The beneficial effects of PPV23 rapidly fade out after inoculation, which is more prominent in old age group. In this sense, PPV23 vaccine is not sufficient in preventing pneumococcal diseases in COPD patients because COPD is the disease of old ages and mortality rate increases exponentially with advancing age. Pneumococcal conjugate vaccine 13 (PCV13) can overcome the waning phenomenon by the production of memory B cells. Although PCV13 is expected to be the best option for the prevention of pneumococcal pneumonia in COPD patients, there are few available studies supporting it.

In this study, we will conduct prospective, multi-center trial with the collaboration of Korean pulmonologists in five university-affiliated hospitals. In this study, we will evaluate influenza and pneumococcal vaccination status, the pathogen distribution, pneumonia severity, and clinical outcomes of hospitalized pneumonia patients with COPD.

If successfully accomplished, this study will enhance the awareness of the preventive use of PCV13 in COPD patients among Korean pulmonologists and, most importantly, it will lead to protection of more COPD patients from pneumococcal pneumonia, one of the most frequent and deadly complication.

DETAILED DESCRIPTION:
1. Objectives; Prospective evaluation of distribution of pathogens and its clinical characteristics in hospitalized pneumonia patients with COPD
2. SUBJECTS AND CENTERS A. Subjects; COPD patients hospitalized for community-acquired pneumonia from Feb, 2017 to Feb, 2018.

   B. Centers; More than five university-affiliated hospitals of Korea
3. OTHER THERAPY; Treatment for COPD with pneumonia will be done by the disposal of attending physicians of each hospital.
4. STUDY DESIGN

   ; prospective, multi-center, cohort study
5. STUDY ANALYSIS A. The required number of COPD patients hospitalized for community-acquired pneumonia

   * The sample size calculations were based on detecting 1 point difference in CURB-65 score between influenza/pneumococcal vaccine recipients and non-recipients (expecting the mean CURB-65 score of 3 points for influenza/pneumococcal vaccine recipients and 4 points for non-recipients), assuming a common standard deviation of 1 point in each group,* a two-tailed test at 5% type I error, and a desired power of 80%. In terms of PCV 13, the estimated sample size for an independent t-test is 90 when we expect that 10% of them were PCV13 recipients and the other 90% were non-recipients (in Korea, 10% of candidates are estimated to be vaccinated with PCV13). Since the CURB-65 scores may not be symmetrically distributed, adding 15% to the required number was considered for a non-parametric test and the desired number of patients with COPD and pneumococcal pneumonia is 104 for the analysis. Total 384 COPD patients admitted for community-acquired pneumonia will be enrolled, assuming 30% prevalence of pneumococcal pneumonia among them (the prevalence of pneumococcal pneumonia is 25~45% in Korea), with allowance of 10% possible data loss.

     * referenced from 'Role of Semi-quantitative Serum Procalcitonin in Assessing Prognosis of Community Acquired Bacterial Pneumonia Compared to PORT PSI, CURB-65 and CRB-65 Journal of Clinical and Diagnostic Research. 2015 Jul, Vol-9(7): OC01-OC04' B. Parameters to be evaluated A) Demographic data . Age, gender, BMI, smoking status, socioeconomic status B) Past medical history

       . Comorbidities; diabetes, hypertension, malignancy, chronic renal disease, chronic liver disease…

       . Smoking status and amount of smoking by pack-year

       . Vaccination status (types and timing)

       - Will be checked both by history taking and by the review of medical record

       - PCV13, PPV23, Influenza vaccine, Zostavax…. C) Diagnostic tests for the identification of pneumonia pathogens

       . Sputum Gram stain/culture (adequacy will be evaluated with the Bartlett criteria)
       * Sputum PCR test for bacterial pneumonia pathogens

         * Multiplex PCR test designed for the detection of S. pneumoniae, M. pneumoniae, L. pneumophila, H. influenza, B. pertussis, C. pneumoniae
       * Urine antigen test(Binax and SS-UAD) for pneumococcus - two aliquots of the urine sample will be frozen and stored for subsequent shipment to the central laboratory (Pfizer Vaccines Research East and Early Development, Pearl River, PA, USA) for Luminex platform-based multiplex UAD assay testing as described previously (Pride et al. Clin Vaccine Immunol 2012;19:1131-41). Processing, storing and shipping of urine samples will be carried out according to Pfizer protocol. Urine will be tested locally using the commercially-available BinaxNOW® S. pneumoniae antigen test also.

         * Control urine samples will be collected from 400 adults without pneumonia according to the Pfizer urine collecting method and stored for subsequent shipment to the central laboratory (Pfizer Vaccines Research East and Early Development, Pearl River, PA, USA) for Luminex platform-based multiplex UAD assay testing.
       * Two sets of blood culture D) Severity scores
       * Pneumonia severity index (PSI)
       * CURB-65 E) Outcome parameters
       * ICU admission rate
       * Mechanical ventilation rate
       * ICU stay and hospital stay
       * Mortality
6. SAFETY;

   ; This is an observational study which evaluates the effects of previously inoculated influenza/pneumococcal vaccine. Treatment for pneumonia and COPD will be done by attending physician with their own disposal. In this setting there would not be ethical issues to be debated.
7. DECISION POINTS/ STATISTICAL METHODS/INTERIM ANALYSIS

   ; The statistics will be purely descriptive. Continuous variables will be presented as mean ± SD or median value with minimum and maximum values. Categorical data will be presented as frequency and percentile. Intergroup comparison of continuous variables will be done with student T test and that of categorical data will be done with Chi-square test or with Fisher's exact test. Statistical significance will be determined at the 5% level. We will consider non-parametric equivalent tests if the distributional assumptions are not suitably made.
8. DATES; Feb 2017 ~ FEB 2018

ELIGIBILITY:
Inclusion Criteria for COPD:

* Currently smoking male or female over 40 years.
* Smoking history ≥ 10 pack-years.
* Post bronchodilator (BD) FEV1/FVC <70% and post BD FEV1 < 80% of predicted.

Exclusion Criteria for COPD

* Chest radiologic abnormalities (taken before the development of pneumonia) which explain the obstructive pattern in pulmonary function.
* Current diagnosis of bronchial asthma.

Inclusion criteria for community-acquired pneumonia

* Newly developed pneumonic infiltrates (lobar-, broncho-, or interstitial-pattern) on chest radiography (taken after the development of respiratory symptoms) with at least 2 of following 3 criteria
* Body temperature (<36℃ or ≥ 38.0℃)
* White blood cell count (<5,000/mm3 or >10,000/mm3)
* Cough and/or sputum

Exclusion Criteria:

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients hospitalized for community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The distribution of pathogens in hospitalized pneumonia patients with COPD | 1 year

SECONDARY OUTCOMES:
Intensive care unit (ICU) admission rate | 1 year
Mechanical ventilation rate | 1 year
The length of ICU stay | 1 year
The length of hospital stay | 1 year
Mortality | 1 year
Age- and gender-matched pneumonia severity | 1 year
  It will be measured by CURB-65 and pneumonia severity index (PSI) in community-acquired pneumonia with COPD

CONTACTS AND LOCATIONS:
Overall Officials: JAE YEOL KIM, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Bundang, Gyeonggi-do
  - Seoul National University, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Chronic obstructive pulmonary disease among adults--United States, 2011. MMWR Morb Mortal Wkly Rep. 2012 Nov 23;61(46):938-43. PMID 23169314
- [Background] Lin SH, Ji BC, Shih YM, Chen CH, Chan PC, Chang YJ, Lin YC, Lin CH. Comorbid pulmonary disease and risk of community-acquired pneumonia in COPD patients. Int J Tuberc Lung Dis. 2013 Dec;17(12):1638-44. doi: 10.5588/ijtld.13.0330. PMID 24200282
- [Background] Rinaudo M, Ferrer M, Terraneo S, De Rosa F, Peralta R, Fernandez-Barat L, Li Bassi G, Torres A. Impact of COPD in the outcome of ICU-acquired pneumonia with and without previous intubation. Chest. 2015 Jun;147(6):1530-1538. doi: 10.1378/chest.14-2005. PMID 25612147
- [Background] Suissa S, Patenaude V, Lapi F, Ernst P. Inhaled corticosteroids in COPD and the risk of serious pneumonia. Thorax. 2013 Nov;68(11):1029-36. doi: 10.1136/thoraxjnl-2012-202872. PMID 24130228
- [Background] Hwang YI, Lee SH, Yoo JH, Jung BH, Yoo KH, Na MJ, Lee JD, Park MJ, Jung CY, Shim JJ, Kim KC, Kim YJ, Choi HS, Choi IS, Lee CT, Lee SD, Kim DJ, Uh ST, Lee HS, Kim YS, Lee KH, Ra SW, Kim HR, Choi SJ, Park IW, Park YB, Park SY, Lee J, Jung KS. History of pneumonia is a strong risk factor for chronic obstructive pulmonary disease (COPD) exacerbation in South Korea: the Epidemiologic review and Prospective Observation of COPD and Health in Korea (EPOCH) study. J Thorac Dis. 2015 Dec;7(12):2203-13. doi: 10.3978/j.issn.2072-1439.2015.12.17. PMID 26793342
- [Background] Myint PK, Lowe D, Stone RA, Buckingham RJ, Roberts CM. U.K. National COPD Resources and Outcomes Project 2008: patients with chronic obstructive pulmonary disease exacerbations who present with radiological pneumonia have worse outcome compared to those with non-pneumonic chronic obstructive pulmonary disease exacerbations. Respiration. 2011;82(4):320-7. doi: 10.1159/000327203. Epub 2011 May 20. PMID 21597277
- [Background] Walters JA, Smith S, Poole P, Granger RH, Wood-Baker R. Injectable vaccines for preventing pneumococcal infection in patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2010 Nov 10;(11):CD001390. doi: 10.1002/14651858.CD001390.pub3. PMID 21069668
- [Background] Almirall J, Bolibar I, Balanzo X, Gonzalez CA. Risk factors for community-acquired pneumonia in adults: a population-based case-control study. Eur Respir J. 1999 Feb;13(2):349-55. doi: 10.1183/09031936.99.13234999. PMID 10065680
- [Background] Lee TA, Weaver FM, Weiss KB. Impact of pneumococcal vaccination on pneumonia rates in patients with COPD and asthma. J Gen Intern Med. 2007 Jan;22(1):62-7. doi: 10.1007/s11606-007-0118-3. PMID 17351841
- [Background] Kweon S, Kim Y, Jang MJ, Kim Y, Kim K, Choi S, Chun C, Khang YH, Oh K. Data resource profile: the Korea National Health and Nutrition Examination Survey (KNHANES). Int J Epidemiol. 2014 Feb;43(1):69-77. doi: 10.1093/ije/dyt228. PMID 24585853